CLINICAL TRIAL: NCT01356927
Title: Etonogestrel Implant or Depot Medroxyprogesterone Acetate for Medication Abortion
Brief Title: Same-day Long-acting Reversible Contraception for Medication Abortion
Acronym: SaLMA
Status: Completed | Type: Observational
Sponsor: Boston University (Other)
Collaborators: Family Planning Fellowship (Other)
Responsible Party: Sponsor
Other Study IDs: H-30255
Record Dates: First submitted 2011-05-18; First posted 2011-05-20 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Abortion; Induced
Keywords: long acting reversible contraception; medical abortion; DMPA; etonogestrel implant; Implanon; contraceptive continuation
MeSH Terms: interventions — N,N-dimethyl-4-anisidine; Medroxyprogesterone Acetate; etonogestrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DMPA: DMPA given at the time of mifepristone for medical abortion
  Interventions: Drug: DMPA
- Etonogestrel implant: Etonogestrel implant placed at the time of mifepristone for medical abortion
  Interventions: Drug: Etonogestrel implant

INTERVENTIONS:
Drug: DMPA — DMPA 150 mg IM given on the day of mifepristone 200 mg po for medical abortion
  Other Names: Depo Provera
  Groups: DMPA
Drug: Etonogestrel implant — Etonogestrel implant placed at the time of mifepristone 200 mg po for medical abortion
  Other Names: Implanon
  Groups: Etonogestrel implant

SUMMARY:
Contraception after abortion is an important public health issue, as women who have an abortion are at high risk for additional unintended pregnancy. In the context of first trimester medical abortion, the standard of care is to administer long-acting reversible contraception, including the etonogestrel implant (Implanon) and depot medroxyprogesterone acetate (DMPA), at a follow-up appointment after the abortion.

The investigators plan to conduct a prospective observational pilot study to evaluate the satisfaction of subjects who have selected either the contraceptive implant or DMPA given on the first day of medical abortion, as opposed to at a follow-up appointment. The investigators will also assess the continuation of DMPA and Implanon at 3, 6, 9, and 12 months after the initial date of administration. In addition, the investigators will assess the total days of bleeding after the abortion, follow-up rate for evaluation of completion of medical abortion, and efficacy of medical abortion.

A total of 40 participants will be recruited, 20 who choose Implanon and 20 who choose DMPA. They will be asked to fill out questionnaires during the course of the study, and will be followed for one year. The study duration including data analysis will be two years.

DETAILED DESCRIPTION:
This is a prospective, observational pilot study of administration of either Implanon or DMPA on the first day of medication abortion. Subjects in this two cohorts will be followed for one year, with questionnaires administered at intake, 2 weeks, 4 weeks, and 3, 6, 9, and 12 months after recruitment.

On the day of recruitment, after the patient has consented both to medication abortion and contraceptive method (Implanon or DMPA), the provider will ask the patient if they are interested in participation in the study. If the patient is interested, a research assistant or investigator will be called to discuss the study in private with the potential subject. Consent will be obtained by the investigator, and the intake questionnaire with baseline contraceptive and demographic data will be administered. Mifepristone for medication abortion will be administered per protocol by the provider, and then Implanon or DMPA will be administered. The clinician who provides the medication abortion will not be the same person as the investigator who is consenting for research. A bleeding diary card will be given to the subject to record daily bleeding. The subject will be requested to return this card by mail in 4 weeks, and will be given an addressed and stamped envelope.

Subjects will be scheduled for a 7-day follow-up appointment as per medication abortion protocol, and at that visit, a short questionnaire regarding the satisfaction with timing of contraceptive method, and number of days of bleeding will be administered. Subjects will then be contacted by their preferred modality (phone, email, or text message) at 2 weeks, to assess for total days of bleeding. If the subject is continuing to have bleeding, they will be contacted again at 4 weeks to assess for total days of bleeding. At each of these contact points, satisfaction with timing of placement, and satisfaction with contraceptive method will be assessed via a Likert scale. Additional contact will be made at 3, 6, 9, and 12 months for all subjects to assess continuation of the contraceptive method.

If unable to contact the subject or listed emergency contacts a total of five times by their preferred or alternate modalities of contact, a letter will be sent along with a self-addressed stamped envelope.

Outcomes (Indicate anticipated primary and any secondary outcomes and how they will be measured):

The primary study objectives are to assess the following:

1. Subject satisfaction with timing of placement as determined by questionnaire
2. Continuation of contraceptive method at 3, 6, 9, and 12 month as determined by questionnaire

The secondary study objectives are to assess the following:

1. Total days of bleeding after the abortion
2. Follow-up rate for evaluation of completion of medication abortion
3. Failure rate of medication abortion
4. The number of women screened for participation
5. Reasons for refusal to participate in the study
6. Reasons for ineligibility
7. The number of women who change their contraceptive method during the year of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Desiring and eligible for medication abortion
* Desiring and eligible for etonogestrel implant or DMPA

Exclusion Criteria:

* Contraindications to DMPA or etonogestrel implant per CDC guidelines regarding United States Medical Eligibility for Contraceptive Use (Centers for Disease Control, 2010)
* Contraindications to mifepristone and misoprostol including ectopic pregnancy, pregnancy with intrauterine device in place, chronic adrenal failure, significant anemia, bleeding disorder, chronic steroid use, inability to follow up, lack of emergency medical access, allergy to mifepristone or misoprostol, malignant liver tumor, benign hepatocellular adenoma, systemic lupus erythematosis with antiphospholipid antibody syndrome, active liver disease, or history of breast cancer or current breast cancer
* Nonworking telephone number (as assessed on initial visit)
* Unable to give informed consent, or unable to speak English, Spanish, or French Creole
* Unable to be contacted because of confidentiality issues
* Currently breastfeeding
* Intending to move away from the Boston area within one year

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will be women who elect a medication abortion at Boston Medical Center and who desire either Implanon or DMPA. Those that appear to meet the eligibility and none of the exclusion criteria will be asked by their clinician if they are interested in participating in the observational study. Those interested will be contacted by the PI or PI's designated staff to discuss details about the study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Satisfaction with timing of contraceptive administration | 7 days, 14 days, 28 days, 3, 6, 9, 12 months
Continuation rate of contraceptive method | 7 days, 14 days, 28 days, 3, 6, 9, 12 months

SECONDARY OUTCOMES:
Number of days of bleeding | 28 days
Follow-up rate after abortion | 14 days
Failure of medical abortion | 7 days
Reasons for non-enrollment | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sarita Sonalkar, MD, Principal Investigator — Boston University
Locations (1):
- Boston University Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sonalkar S, McClusky J, Hou MY, Borgatta L. Administration of depot medroxyprogesterone acetate on the day of mifepristone for medical abortion: a pilot study. Contraception. 2015 Feb;91(2):174-7. doi: 10.1016/j.contraception.2014.10.010. Epub 2014 Nov 6. PMID 25481376
- [Derived] Sonalkar S, Hou MY, Borgatta L. Administration of the etonogestrel contraceptive implant on the day of mifepristone for medical abortion: a pilot study. Contraception. 2013 Nov;88(5):671-3. doi: 10.1016/j.contraception.2013.07.008. Epub 2013 Jul 29. PMID 24028749